CLINICAL TRIAL: NCT07404735
Title: A Randomized, Open-label and Parallel Study to Evaluate the Pharmacokinetics and Safety of CKD-846 in Healthy Male Subjects
Brief Title: A Clinical Trial to Compare and Evaluate Evaluate the Pharmacokinetics and Safety of CKD-846
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A133_02PK2504
Record Dates: First submitted 2026-01-29; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Benign Prostate Hypertrophy(BPH)
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- A1 (Test group) (Experimental): CKD-846, Single dose
  Interventions: Drug: CKD-846
- A2 (Test group) (Experimental): CKD-846, Single dose
  Interventions: Drug: CKD-846
- A3 (Test group) (Experimental): CKD-846, Single dose
  Interventions: Drug: CKD-846
- R (Reference group) (Experimental): D091, Multi dose
  Interventions: Drug: D091

INTERVENTIONS:
Drug: CKD-846 — once administration of Investigational Product
  Arms: A1 (Test group); A2 (Test group); A3 (Test group)
Drug: D091 — once administration of Investigational Product
  Arms: R (Reference group)

SUMMARY:
A Clinical trial to compare and evaluate evaluate the pharmacokinetics and safety of CKD-846

DETAILED DESCRIPTION:
A randomized, open-label and parallel study to evaluate the pharmacokinetics and safety of CKD-846 in healthy male subjects

ELIGIBILITY:
Inclusion Criteria:

1. Healthy man aged between 19 to 55 at screening
2. Weight ≥ 55kg
3. Body mass index (BMI) of 18.5 to 27.0kg/m2
4. Those who agree to contraception from the first Investigational Product(IP) dosing day till 6 months after the last dosing day and decide not to provide sperm during the participation of clinical trial
5. Those who voluntarily decide to participate in paper and agree to comply with the cautions after fully understand the detailed description of this clinical trial

Exclusion Criteria:

1. Those who have clinically significant disease or medical history of Hepatopathy, Renal, Neurological, Immunity, Respiratory, Endocrine, urinary, tumor or Psychical disorder
2. Those who have a history of clinically significant cardiovascular diseases such as myocardial infarction, angina pectoris, ventricular arrhythmia, heart failure, left ventricular outflow tract stenosis, stroke, and transient ischemic attack within 2 years prior to the first administration of the investigational drug
3. Those with eye diseases including genetic degenerative retinal diseases, including retinitis pigmentosa
4. Those with a past history of erection lasting more than 4 hours and priapism while taking PDE5 inhibitors such as tadalafil
5. Those who have a history of gastrointestinal surgery except simple appendectomy and hernia surgery which can interfere with drug absorption
6. Persons with a history of clinically significant hypersensitivity to drugs or additives, including ingredients of clinical investigational drugs
7. Those who have genetic problems such as galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption
8. A person who is judged to be unsuitable as a test subject in a screening test conducted within 28 days before administration of the investigational drug
9. Those who has a drug abuse history within one year or positive reaction on urine drug screening test.
10. Those who has taken over-the-counter or prescription drugs, excluding topical agents without significant systemic absorption, within a specified period of time and the administered drug is judged to have an effect on this test or may affect the safety of the subject
11. People who need to take nitrate preparations or nitric oxide donors etc. regularly or intermittently during the clinical trial period
12. Those who continuously smoke excessively or consume caffeine or alcohol
13. A person who consumed food containing grapefruit within 7 days before the first administration of the investigational drug
14. Persons who participated in another clinical trial (including bioequivalence test) and received an investigational drug within 180days prior to the date of first administration of the investigational drug
15. Those who donated whole blood within 60 days before the first date of administration and donated ingredients within 30 days
16. Those who have received blood transfusion in 30 days
17. Those who are deemed insufficient to participate in clinical study by investigators

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male
Enrollment: 32 (Estimated)
Dates: Start 2026-02-23 (Estimated); Primary Completion 2026-05-27 (Estimated); Study Completion 2026-06-02 (Estimated)

PRIMARY OUTCOMES:
Plasma Concentration of D091 | Pre-dose, Post-dose Day1~Day34 (During the administration period)
  Concentration of During the administration period
Plasma Concentration of CKD-846 | Pre-dose, Post-dose Day1~Day91 (During the administration period)
  Concentration of During the administration period

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No